CLINICAL TRIAL: NCT02777047
Title: Coordination of Oral Anticoagulant Care at Hospital Discharge (COACHeD): A Pilot Randomized Trial
Brief Title: Coordination of Oral Anticoagulant Care at Hospital Discharge
Acronym: COACHeD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Collaborators: Hamilton Academic Health Sciences Organization (Other); Institute for Safe Medication Practices Canada (Unknown); Canadian Institutes of Health Research (CIHR) (Other Government); Hamilton Health Sciences Corporation (Other); Brant Community Healthcare System (Unknown); Grand River Hospital (Other); Niagara Health System (Other)
Responsible Party: Principal Investigator, Dr. Anne Holbrook, Director, Division of Pharmacology and Toxicology, St. Joseph's Healthcare Hamilton
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Anticoag Safety
Record Dates: First submitted 2016-05-13; First posted 2016-05-19 (Estimated); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Anticoagulants
Keywords: Thromboembolism; Medication Safety; Hospital-community collaboration; Pilot RCT; Telehealth
MeSH Terms: conditions — Thromboembolism

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The interdisciplinary multimodal intervention is led by a clinical pharmacologist and includes: a detailed discharge medication reconciliation and management plan focused on oral anticoagulants at hospital discharge; a circle of care handover and coordination with patient, hospital team and community providers; and early post-discharge follow-up virtual medication check-up visits at 24 hours, 1 week, and 1 month.
  Interventions: Other: Anticoagulation Coordinated Care
- Control (No Intervention): Patients allocated to the control group will receive usual care, plus the URL to Thrombosis Canada website. Usual care in the participating sites includes OAC management by family doctors except for new thromboembolic events which will be followed short term by thromboembolism or hematology specialists, complicated atrial fibrillation which will have cardiology involved temporarily, and a small proportion of warfarin management which is provided in an anticoagulation clinic. This choice of control group is the most relevant for generalizability to both academic and community practices.

INTERVENTIONS:
Other: Anticoagulation Coordinated Care — see above
  Arms: Intervention

SUMMARY:
Oral anticoagulants (OACs - warfarin, dabigatran, rivaroxaban, apixaban and edoxaban) are the very top cause of serious drug-related harm. More than 7 million prescriptions are dispensed annually for oral anticoagulants (OAC) in Canada, with more than 340,000 elderly recipients in the Ontario Drug Benefit Program alone. Because of their very high and chronic utilization, their large benefit in lowering important clinical events (stroke, clots, death) and their high potential for major harm (primarily bleeds, which can be fatal), OACs are the highest priority for improving medication safe and effective use. The early period after hospital discharge is clearly high risk, with three times the usual rate of major bleeds compared with later.

Patients and families frequently note confusion about their medications after leaving the hospital due to errors or lack of detailed communication to their health care team at the time of discharge. The confusion, errors, and lack of communication are highly associated with lack of adherence to medications and resulting worse health outcomes. The combination of waste of medication and bad outcomes that result from medication errors, are estimated to cost our health care system several billion dollars annually. Since our leading economists are declaring health care to be unsustainable in its current delivery forms, it is time to find and evaluate more cost-effective ways to improve anticoagulation safety. The investigators will do this by structuring discharge medication assessment, with more expert management, formal written and verbal handovers to the patients, their family and their hospital and community doctors, pharmacists and home care; follow-up by virtual visits after discharge, and coordinate advice and communication to extend access to and reduce the cost of expert guidance. The investigators expect that this intervention will decrease anticoagulant-related adverse events and improve ratings of the coordination of care. If this occurs, the investigators will develop a business plan for regions, provinces and territories to scale up the intervention to a national level.

DETAILED DESCRIPTION:
Design: Randomized controlled pilot trial, two parallel groups, blinded outcome assessment.

Eligibility Criteria: Inclusion criteria include a) adult patients within a day of their hospital discharge from internal medicine services with a discharge prescription for an OAC intended to be taken for at least 4 weeks, b) discharge is to home or to a congregant setting such as retirement home where the patient manages their own medications, c) English-speaking and d) capable of providing informed consent. Ability to consent will be measured by the COACHeD Capacity to Consent test, requiring a score of 14 or more. If the patient does not pass, a close caregiver (defined as a family member in daily contact with the patient and involved in their medication supervision), will be invited to provide consent on the patient's behalf by signing a caregiver consent form.

Patients will be excluded if they are less than 18 years of age, have an expected lifespan of less than 3 months, will be discharged to long term care or other institution where medications are controlled by staff, or decline informed consent.

Intervention: Intervention patients will receive:

1. Interdisciplinary intervention led by a clinical pharmacologist who is a leader in evidence-based prescribing - includes a detailed discharge medication reconciliation and management plan focussed on oral anticoagulants at hospital discharge; a circle of care handover and coordination with patient, hospital team and community providers; three scheduled early post-discharge virtual medication check-up visits at 24 hours, 1 week, and 1 month with triage of any problems. Medication reconciliation is a process mandated by national accreditation bodies, with incomplete and variable uptake, which reviews hospital-administered medications compared to pre-admission medications. Medication management is the more complex task of assessing and revising medications in light of patient diagnoses, current symptoms and signs, risk factors, allergies and intolerances, other medications, goals, etc. In this study, all medications will be reviewd with a focus on OAC choice, dosage, indication, duration, potential drug interactions, patient risk factors for thromboembolism versus bleeding, drug insurance, adherence challenges and health literacy. A study pharmacist with additional training, will complete the detailed medication reconciliation.
2. Hand-overs to the community care team including the main patient caregiver (if applicable), family physician, medical specialist(s), and community pharmacist, using a templated consult summary including an OAC Monitoring Checklist (example consult note shown in Figure 2). The monitoring is based on: a) best evidence (updated guidelines and dedicated evidence review using the CLOT repository of CanVECTOR and McMaster's Health Information Research Unit), and decision aid content for patients and their families to assist in anticoagulant knowledge and adherence, b) best practices regarding discharge medication management, virtual care, scalable coordination of care with clear accountability, communication and teletriage where situations require medical intervention. All consult notes are reviewed in detail with the Clinical Pharmacologist.
3. 'Virtual visits' (secure video calls from within our electronic medical record (EMR) or phone visits where video is not possible) by the study pharmacist at three follow-up time points - 24 hours post-discharge to ensure the discharge prescription medications were obtained and understood, OAC Monitoring Checklist, review other medications, solicit concerns; and at 1 week and 1 month to ensure medication adherence, review the OAC Monitoring Checklist and other medications, and solicit concerns. After each follow-up visit, a summary consult note will be sent to all circle of care providers, and any clinical events or serious concerns will be addressed by the Clinical Pharmacologist or directed to patient's family physician via phone call or direct email. Each follow-up visit with intervention patients will be recorded and tracked to ensure adherence to protocols.
4. Teletriage- The patients have the study pharmacist's contact information and can phone for assistance at any time. The study pharmacist is in constant communication with a Clinical Pharmacologist investigator for guidance. An expert Thrombosis specialist will be available on call as needed.

ELIGIBILITY:
Inclusion criteria include a) adult patients within a day of their hospital discharge from internal medicine services with a discharge prescription for an OAC intended to be taken for at least 4 weeks, b) discharge is to home or to a congregant setting such as retirement home where the patient manages their own medications, c) English-speaking and d) capable of providing informed consent. Ability to consent will be measured by the COACHeD Capacity to Consent test, requiring a score of 14 or more. If the patient does not pass, a close caregiver (defined as a family member in daily contact with the patient and involved in their medication supervision), will be invited to provide consent on the patient's behalf by signing a caregiver consent form.

Patients will be excluded if they are less than 18 years of age, have an expected lifespan of less than 3 months, will be discharged to long term care or other institution where medications are controlled by staff, or decline informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2020-12-16 (Actual); Primary Completion 2022-06-27 (Actual); Study Completion 2022-06-27 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | 1 year
  Feasibility assessments are used to determine whether a research study is likely to be delivered successfully, taking into account the practical aspects of managing the project such as recruitment rate
Participant retention rate | 3 months
  Feasibility assessments are used to determine whether a research study is likely to be delivered successfully, taking into account the practical aspects of managing the project such as participant retention rate
Estimated resources required per patient to complete the main trial | 3 months
  Feasibility assessments are used to determine whether a research study is likely to be delivered successfully, taking into account the practical aspects of managing the project such as resources required per patient to complete participation in the trial.

SECONDARY OUTCOMES:
Adverse Anticoagulant Safety Events composite (AASE) | 3 months
  Any of thromboembolic events or clinically relevant bleeding or death. Thromboembolic events include objectively verified ischemic stroke, systemic embolism, pulmonary embolism, or DVT. Clinically relevant bleeds in this study is defined as bleeding that causes death, hospitalization or Emergency Department visits.
Coordination and Continuity of Care Questionnaire | 3 months
  Adapted from Health Quality Ontario's draft guidance and a Rand instrument, the Coordination and Continuity of Care Questionnaire is designed to measure the quality of the transitional and follow-up care.
Patient Quality of Life | 3 months
  The EQ-5D-5L is the 5-level classification system of the EQ-5D, a measure of health status from the EuroQol Group. Using EQ-5D-5L, respondents are asked a short series of questions about mobility, self-care, usual activities, pain discomfort, and anxiety/ depression, as well as a summary visual analogue scale. This scale, which provides utility measurements, has been well validated for the Canadian population.
Patient Knowledge of OAC Management | 3 months
  Insufficient patient knowledge about OAC may predict poor medication adherence and inadequate anticoagulation control. The COACHeD OAC Knowledge Questionnaire tests knowledge of the therapeutic objective, process of use, safety and maintenance of the medications.
Satisfaction with Care | 3 months
  Satisfaction reported by patients and by key health professionals is one of the recommended outcomes to report in medical research, as it may influence adherence. This outcome will be assessed by the Patient/Caregiver Study Satisfaction Survey and by the Provider Study Satisfaction Survey.
Medication Problems | 3 months
  We will be assessing problems with appropriateness, with medication errors characterized using the NCC-MERP scale and with medication adherence and attitudes as measured by COMPETE Medication Problems Questionnaire.
Resource Utilization | 3 months
  This is a key outcome to determine cost-effectiveness and cost-utility which then determines whether health care systems might pay for this type of care. We will be measuring all types of health care utilization by patients.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Holbrook, MD,PharmD,MSc, Principal Investigator — Director, Clinical Pharmacology & Toxicology
Locations (1):
- St Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Holbrook A, Troyan S, Telford V, Koubaesh Y, Vidug K, Yoo L, Deng J, Lohit S, Giilck S, Ahmed A, Talman M, Leonard B, Refaei M, Tarride JE, Schulman S, Douketis J, Thabane L, Hyland S, Ho JM, Siegal D. Coordination of oral anticoagulant care at hospital discharge (COACHeD): pilot randomised controlled trial. BMJ Open. 2024 May 1;14(5):e079353. doi: 10.1136/bmjopen-2023-079353. PMID 38692712
- [Derived] Holbrook AM, Vidug K, Yoo L, Troyan S, Schulman S, Douketis J, Thabane L, Giilck S, Koubaesh Y, Hyland S, Keshavjee K, Ho J, Tarride JE, Ahmed A, Talman M, Leonard B, Ahmed K, Refaei M, Siegal DM. Coordination of Oral Anticoagulant Care at Hospital Discharge (COACHeD): protocol for a pilot randomised controlled trial. Pilot Feasibility Stud. 2022 Aug 2;8(1):166. doi: 10.1186/s40814-022-01130-z. PMID 35918731
- [Derived] Benipal H, Holbrook A, Paterson JM, Douketis J, Foster G, Thabane L. Predictors of oral anticoagulant-associated adverse events in seniors transitioning from hospital to home: a retrospective cohort study protocol. BMJ Open. 2020 Sep 22;10(9):e036537. doi: 10.1136/bmjopen-2019-036537. PMID 32963065